CLINICAL TRIAL: NCT06495970
Title: Pulmonary Artery DenerVation Clinical Study Using the Gradient Denervation System in Heart Failure Patients With Pulmonary Hypertension Group 2 (PreVail-PH2 OUS Study)
Acronym: PreVailPH2 OUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gradient Denervation Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-003
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PADN with Gradient Denervation System (Experimental)
  Interventions: Device: Gradient Denervation System

INTERVENTIONS:
Device: Gradient Denervation System — The Gradient Denervation System delivers ultrasound ablation to planned locations in the pulmonary artery to down-regulate the sympathetic nervous drive. The system includes a sterile, single-use catheter that is designed to centrally position the transducer within the arterial target zone for consistency of ablation.

SUMMARY:
Characterize the impact of pulmonary artery denervation on the quality of life in Heart Failure Patients with Group 2 Pulmonary Hypertension

DETAILED DESCRIPTION:
The Gradient Denervation System delivers ultrasound ablation to planned locations in the pulmonary artery to down-regulate the sympathetic nervous drive. The system includes a sterile, single-use catheter that is designed to centrally position the transducer within the arterial target zone for consistency of ablation.

ELIGIBILITY:
Inclusion Criteria:

* Mean Pulmonary Artery Pressure (mPAP) >20 mmHg at rest
* Pulmonary Vascular Resistance (PVR) ≥ 3WU at rest
* Pulmonary Capillary Wedge Pressure > 15 mmHg (at rest) or > 18 with passive leg raise
* NYHA Class II or III
* Glomerular Filtration Rate (GFR) ≥ 25 ml/min

Exclusion Criteria:

* Unwilling to provide informed consent or complete follow-up assessments
* Life expectancy of < 2 years
* Inability to take dual antiplatelet or anticoagulants, hypersensitivity or allergy to aspirin or clopidogrel
* Unable to tolerate right heart catheterization
* Severe aortic, mitral or pulmonary valve regurgitation
* Clot or Thrombus in any potential target ablation zone (right, left or main pulmonary artery)
* Systemic infection or localized infection/rash at planned access site at time of procedure
* CRT, ICD, Pacemaker or other Interventional cardiac procedure (except RHC) within the last 3 months

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Device related serious adverse events | 30-days post-treatment
  Frequency of device related SAEs

SECONDARY OUTCOMES:
Mean change from baseline in Pulmonary Vascular Resistance (woods units) | 6 month post-treatment
  Calculated percent mean change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Julie Etheridge, Study Director — Gradient
Locations (3):
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No